CLINICAL TRIAL: NCT02953496
Title: A Phase 1 Multi-Center, Dose-Escalation Study of Vonapanitase Administered Percutaneously to the Superficial Femoral or Popliteal Artery in Patients With Peripheral Artery Disease
Brief Title: Safety/ Feasibility of Percutaneous Administration of Vonapanitase as Monotherapy for Peripheral Artery Disease (PAD) of the SFA and Popliteal Arteries
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in operating plans
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-201-110
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; PAD; vonapanitase; claudication; superficial femoral artery; SFA; popliteal artery; stenosis; elastase; chymotrypsin-like elastase 1; CELA1; PRT-201
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Constriction, Pathologic | interventions — cholesterol-binding protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vonapanitase (Experimental)
  Interventions: Drug: vonapanitase

INTERVENTIONS:
Drug: vonapanitase — Vonapanitase will be administered to the target lesion of the SFA or PA via percutaneous needle injection under ultrasound guidance.
  Other Names: PRT-201

SUMMARY:
The research study is designed to assess the technical feasibility and safety of percutaneous administration of vonapanitase to the superficial femoral or popliteal artery in patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Clinical diagnosis of PAD secondary to atherosclerosis affecting a lower limb.
3. ABI <0.90 at rest or with exercise, or a toe-brachial index (TBI) <0.70 if ABI value is >1.30 (non-compressible), or radiographic evidence of PAD that correlates with clinical symptoms.
4. Rutherford category 2-4.
5. Screening duplex Doppler ultrasound with a SFA or PA lesion with a PSVR >2.4.
6. De novo lesion, not previously treated by angioplasty, atherectomy, or stent.
7. If female and of childbearing potential (premenopausal and not surgically sterile) must have a negative pregnancy test at the screening visit and be willing to use contraception from the time of the screening visit to 1 week following study drug administration. Acceptable methods of birth control include abstinence, barrier methods with spermicide, implants, injectables, oral contraceptives, intra-uterine device, or a vasectomized partner.
8. Ability to understand and comply with the requirements of the entire study and communicate with the study team.
9. Ability to provide written informed consent using a document that has been approved by the required institutional review board.

Exclusion Criteria

1. Patients in whom arterial insufficiency in the lower extremity is the result of an immunologic or inflammatory non-atherosclerotic disorder (e.g., Buerger's disease, vasculitis).
2. Total occlusion of the SFA or PA in the index leg.
3. Planned surgical or endovascular procedures to the affected leg on the day of or within 28 days of study drug administration.
4. Deep vein thrombosis within the past 3 months.
5. Known bleeding disorder.
6. Presence of any arterial aneurysm in the index leg.
7. Known hypercoagulable state (e.g., protein C deficiency, factor V Leiden mutation, prothrombin G20210A mutation).
8. Platelet count <130K, hematocrit <30%, bilirubin or ALT >3.0 times the upper limit of normal.
9. Arterial systolic BP >200 mmHg or diastolic BP >100 mmHg at screening or day of procedure.
10. Pregnancy, lactation or plans to become pregnant during the course of the study.
11. Presence of any significant medical condition that might significantly confound the collection of safety and efficacy data in this study.
12. Malignancy or treatment for malignancy within the previous 12 months with the exception localized basal cell or squamous cell skin cancer, or any cancer in situ.
13. Treatment with any investigational drug within the previous 30 days or investigational antibody therapy within 90 days prior to signing informed consent.
14. Known allergy to contrast media, iodine, lidocaine, prilocaine, or EMLA Cream (lidocaine 2.5% and prilocaine 2.5%).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months following study drug administration
  Safety assessments include physical exams, duplex Doppler ultrasound and routine serum chemistry and hematology tests
Technical success of percutaneous injection | Intraprocedural
  Technical success of study drug administration will be assessed by the extent of circumferential and longitudinal coverage of the artery using a protocol-defined assessment scale

OTHER OUTCOMES:
Peak systolic velocity ratio [PSVR] | 14 days and 6 months following study drug administration
Minimum lumen diameter [MLD] | 14 days and 6 months following study drug administration
Rutherford category | 14 and 28 days, and 6 months following study drug administration
Ankle-brachial index [ABI] | 14 days and 6 months following study drug administration
6-minute walk test [6MWT] | 14 days and 6 months following study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States